CLINICAL TRIAL: NCT04209140
Title: Optimizing Response to Li Treatment Through Personalized Evaluation of Individuals With Bipolar I Disorder: The R-LiNK Initiative
Acronym: R-LiNK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P180101; 2018-002263-26 (EudraCT Number)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Bipolar I Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- bipolar I disorders who initiate lithium treatment
  Interventions: Drug: lithium treatment

INTERVENTIONS:
Drug: lithium treatment — Decisions relating to treatment are also considered the clinician's responsibility to be made according to bipolar treatment guidelines and international standards of care (e.g. discontinuation, co-prescriptions, and according to SmPC in force). After the clinician has confirmed the indication of Lithium treatment as well as the absence of contra-indicated concomintant medication (NSAIDs and Diuretics) and after pre-
  Lithium evaluations confirm the absence of contra-indication, Lithium is initiated following standard of care:
  progressive titration to reach therapeutic plasma levels. Clinicians will use the therapeutic range provided by the laboratory they use in their usual clinical practice and according to the type of Lithium they prescribe.

SUMMARY:
Bipolar disorder (BD), especially BD type I, is a highly prevalent mental disorder and a is a highly prevalent mental disorder and an important factor for suicide. Lithium is the key treatment for prevention of BD relapse and has a proven suicide prevention effect. Whilst many cases become asymptomatic with lithium treatment, the majority show sub-optimal response.

The objectives of this project are to:

* improve outcomes of bipolar I disorder (BDI) cases prescribed lithium through the application of stratified approaches
* optimize the early prediction of lithium response using a set of multi-modal biomarkers ("blood omics", Magnetic Resonance Imaging and Li7-Magnetic Resonance Spectroscopy derived-markers)
* develop a multidisciplinary multinational network of experts to undertake this and future projects on personalized diagnostics and therapeutics and
* implement new, powerful technologies to characterize brain lithium distribution and the blood molecular signature of lithium in responders and non-responders.

This cutting edge approach will identify the eligibility criteria for treatment with lithium in BD in terms of response, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Decision to prescribe Li as a prophylactic treatment based on clinicians' assessment
* Confirmed diagnosis of BD1 according to DSM-5 criteria
* Aged 18-70 years.
* Able and willing to give written informed consent
* consents to blood sample for the purpose of the RLiNK study
* Covered by a Social Security Insurance where applicable
* Patients on Curatorship (consent form signed by the patient and specific consent form for the curator)

Exclusion Criteria:

* Trial of Lithium undertaken within the last 6 months
* Lifetime history of mood disorder better explained by a DSM-5 definition for schizoaffective disorder
* Pre-lithium screening suggest that Lithium initiation is contraindicated:
* Incompatible concurrent treatments: long-term use of non- steroidal anti-inflammatory drug or diuretics for a known and established comorbid disorder with no possible alternative treatment (i.e. absolute contra-indication to Li treatment)
* Health issues (risk of worsening of a pre-existing condition) Psoriasis, Brugada syndrome
* Renal dysfunction: Glomerular Filtration rate below 60mL/min/1.73m 2
* On-going Pregnancy or planned pregnancy on the next 2 years
* Lactating and breast feeding women (see SmPc)
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with bipolar I disorder
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Responder | month 24
  Good Responder The individual meets criteria for sustained remission, namely they experience euthymia (defined as a score on the Quick Inventory of Depressive Symptoms (qIDS)<6 and the Bech Rafaelson Mania Scale (BRMS)<7) for at least 8 weeks during the two-year follow-up period without evidence of relapse into a syndromal episode of BD at any time after achieving sustained euthymia. AND No addition of a new mood stabilizer with the purpose of promoting mood stabilisation after lithium initiation
  Non Responder
  The individual:
  Fails to meet criteria for sustained remission (euthymia defined as a score on the qIDS<6 and the BRMS<7 for a minimum period >=8 consecutive weeks) during the two-year follow-up.
  OR Experiences >=1 relapse into a syndromal episode of BD of any polarity during the two-year follow-up period without any period of sustained remission
  Definition of a Partial Responder All cases not fulfilling the criteria of Good Responders or Non Responders

SECONDARY OUTCOMES:
Adherence | Month 24
  Adequate adherence will be defined as the individual taking at least 70% of the Li prescribed (i.e. either >70% prescribed dose &/or >70% of the time) based on the monthly assessment of adherence
Alda Scale | Month 24
  Alda scale defined in the following article : Grof P, Duffy A, Cavazzoni P, Grof E et al. Is response to prophylactic lithium a familial trait? J Clin Psychiatry. 2002 Oct;63(10):942-7.
Responder - sensitivity | Month 24
  Good Responders= Recorded improvement of illness activity is >=70% AND no addition of mood stab after Li initiation Non Responders= Recorded improvement of illness activity is <=30% whatever the treatment has been Partial Responders = Recorded improvement of illness activity is between 70 and 30% whatever the treatment has been OR Recorded improvement of illness activity is >=70% but the addition of mood stab after Li initiation has occurred
Time to new BD | Month 24
  Time to a new Bipolar Disorder (BD) episode, defined as the delay between inclusion and the date of the diagnosis of new Bipolar disorder
Time to BD hospitalization | Month 24
  Time to a new hospitalization for BD, defined as the delay between inclusion and the date of new hospitalization for Bipolar disorder
Time to new mood stabilizer | Month 24
  Time to prescription of a new mood stabilizer, defined as the delay between inclusion and the date of prescription of a new mood stabilizer
Monthly qIDS | monthly from month 1 to month 24
  Quick Inventory of Depressive Symptoms (qIDS)
Monthly BRMS | monthly from month 1 to month 24
  Bech Rafaelson Mania Scale (BRMS)
Monthly BPRS | monthly from month 1 to month 24
  Brief Psychosis Rating Scale (BPRS)
Monthly ISS | monthly from month 1 to month 24
  Internal State Scale (ISS)
Monthly LIFE-II | monthly from month 1 to month 24
  Longitudinal Interval Follow-up Evaluation (LIFE-II)
WHODAS | Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, month 24
  World Health Organisation Disability Assessment Scale (WHODAS)
Cost-effectiveness | Month 24
  EuroQOL-5D scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fernand Widal, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided